CLINICAL TRIAL: NCT04363515
Title: Pilot Social Support Counseling Intervention for Kidney Transplant Candidates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HSR 19-4710
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Results first posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Kidney Transplant
Keywords: Interventional Counseling; Kidney Transplant; Interventional Mapping; Counseling; Social Support Networks; Dialysis

STUDY DESIGN:
Intervention Model Description: A control group versus interventional group. Interventional group and their social support network will complete questionnaire.
Who Masked: Outcomes Assessor
Masking Description: This is a pilot feasibility study, but statisticians will be blinded to group assignment when assessing outcomes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Pre-Transplant Counseling Intervention (No Intervention): Subjects in the control arm will undergo usual pre-transplant counseling as per the standard of care.
- Social Support Network Counseling Intervention (Experimental): Subjects in the intervention arm will undergo an additional pretransplant counseling session along with members of their social support networks between 2-12 weeks after their initial transplant evaluation and counseling
  Interventions: Behavioral: Social support network counseling intervention

INTERVENTIONS:
Behavioral: Social support network counseling intervention — Pilot social support counseling intervention for kidney transplant candidates along with their social support networks
  Arms: Social Support Network Counseling Intervention

SUMMARY:
Feasibility pilot social support counseling intervention for kidney transplant candidates

DETAILED DESCRIPTION:
Individuals who are eligible for kidney transplant will be randomized into two groups, control and interventional counseling. The control group will be given a simple survey to fill and return while the interventional counseling will go through a second counseling session along with members of their social support networks. The interventional counseling will then complete the survey (same as control group). Survey answers will be recorded within REDCAP.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 18-80
* Being considered for kidney transplant
* Part of social support network for an individual being considered for kidney transplant.
* Physically and Mentally able to participate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hennepin Healthcare Research Institute, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided
There might be an exchange of data with our collaborators with the study at the University of Minnesota-Twin Cities

REFERENCES:
- See also: American Transplant Congress oral abstract — https://atcmeetingabstracts.com/abstract/journey-to-transplant-a-pilot-feasibility-trial-of-a-virtual-counseling-intervention-for-patients-and-their-social-support-networks-to-improve-access-to-kidney-transplant/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants for the feasibility pilot trial were recruited from two transplant centers in Minnesota, Hennepin Healthcare and The University of Minnesota, between August 2020 and March 2021.
Period: Overall Study
Arm/Group | Usual Pre-Transplant Counseling Intervention | Social Support Network Counseling Intervention
Started | 8 | 15
Completed | 8 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Pre-Transplant Counseling Intervention | Social Support Network Counseling Intervention | Total
Number analyzed (Participants) | 8 | 15 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (12.6) | 60 (11.3) | 60 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 4 | 10 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 6 | 3 | 9
  Asian American | 1 | 0 | 1
  Latinx | 0 | 1 | 1
  White | 1 | 11 | 12
  Other | 0 | 0 | 0
Education [Count of Participants; unit: Participants]
  Some High School | 1 | 2 | 3
  High School Diploma | 3 | 3 | 6
  Some College or Higher | 4 | 10 | 14
Income [Count of Participants; unit: Participants]
  < $15,000 | 2 | 2 | 4
  $15,000-30,000 | 2 | 2 | 4
  $30,000-45,000 | 1 | 3 | 4
  $45,0000-60,000 | 0 | 1 | 1
  $60,000-75,000 | 1 | 1 | 2
  >$75,000 | 0 | 5 | 5
  Choose not to answer | 2 | 1 | 3
Employment [Count of Participants; unit: Participants]
  Retired | 4 | 6 | 10
  Unemployed | 1 | 4 | 5
  Full-Time Homemaker | 1 | 0 | 1
  Employed Full Time | 1 | 3 | 4
  Employed Part Time | 1 | 1 | 2
  Unable to Work | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Correct Answers on Knowledge of Kidney Transplant Options Assessment
Description: Question key (true/false, multiple choice)
  1. A patient on dialysis has the same level of kidney functioning as a patient with a transplanted kidney.
  2. In general, patients can live at least 5 years longer with a kidney transplant than if they stayed on dialysis.
  3. In general, most people on dialysis are happier with the quality of their lives than people with transplants.
  4. Patients have better health outcomes if they receive a transplant before starting dialysis.
  5. If a patient waits long enough on the waitlist, a matching kidney from someone who has died will definitely become available.
  6. About what percentage of all transplanted kidneys function for at least one year?
  7. Nationally, how long do patients generally wait on the waitlist for a kidney from someone who has died?
  8. Compared to transplants from donors who have died, how long do transplants from living donors last?
  9. What is the chance that a living donor or recipient would die undergoing surgery?
Time Frame: one month
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Pre-Transplant Counseling Intervention | Social Support Network Counseling Intervention
Number analyzed (Participants) | 8 | 15
Participants
  Question 1: Answered Correctly | 6 | 14
  Question 1: Answered Incorrectly | 2 | 1
  Question 2: Answered Correctly | 8 | 15
  Question 2: Answered Incorrectly | 0 | 0
  Question 3: Answered Correctly | 6 | 13
  Question 3: Answered Incorrectly | 2 | 2
  Question 4: Answered Correctly | 3 | 9
  Question 4: Answered Incorrectly | 5 | 6
  Question 5: Answered Correctly | 0 | 9
  Question 5: Answered Incorrectly | 8 | 6
  Question 6: Answered Correctly | 0 | 10
  Question 6: Answered Incorrectly | 8 | 5
  Question 7: Answered Correctly | 4 | 6
  Question 7: Answered Incorrectly | 4 | 9
  Question 8: Answered Correctly | 2 | 10
  Question 8: Answered Incorrectly | 6 | 5
  Question 9: Answered Correctly | 1 | 11
  Question 9: Answered Incorrectly | 7 | 4

2. Secondary Outcome: Difference in Decisional Conflict Scores
Description: questionnaire (Ottawa Decisional Conflict scale)
Time Frame: one month
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Pre-Transplant Counseling Intervention | Social Support Network Counseling Intervention
Number analyzed (Participants) | 8 | 15
Participants
  Do you feel sure about the best choice for you?: Yes | 7 | 14
  Do you feel sure about the best choice for you?: No | 1 | 1
  Do you know the benefits and risks of getting a kidney transplant?: Yes | 4 | 15
  Do you know the benefits and risks of getting a kidney transplant?: No | 4 | 0
  Are you clear about which benefits and risks matter most to you?: Yes | 6 | 15
  Are you clear about which benefits and risks matter most to you?: No | 2 | 0
  Do you have enough support and advice to make a choice?: Yes | 6 | 15
  Do you have enough support and advice to make a choice?: No | 2 | 0

ADVERSE EVENTS:
Time Frame: No adverse event data were collected.
Description: No mortality, serious, or other adverse events were monitored or assessed.
Arm/Group | Usual Pre-Transplant Counseling Intervention | Social Support Network Counseling Intervention
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-10-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT04363515/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT04363515/SAP_001.pdf